CLINICAL TRIAL: NCT03652285
Title: Universal Partially Covered Removable Self-Expanding Stent and Anchoring System for the Treatment of Refractory Benign Esophageal Strictures (UAS-RBS): a Safety Study
Brief Title: UAS-RBS: a Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2017/543
Record Dates: First submitted 2018-07-10; First posted 2018-08-29 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Refractory Benign Strictures

STUDY DESIGN:
Intervention Model Description: As a proof of concept, feasibility study - First In Man Study (FIM). The study will enroll 10 patients and an additional 10% of patients to compensate for potential attrition during follow-up, resulting in a sample size of 11 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal stent implantation (UAS-RBS implantation) (Experimental): Esophageal stent implantation (UAS-RBS implantation) at J0, removal after 6 months and follow-up for 6 months
  Interventions: Device: Esophageal stent implantation; Device: Stent removal

INTERVENTIONS:
Device: Esophageal stent implantation — An upper endoscopy will be performed with the use of fluoroscopy. Depending on the size of the stricture a dilation can be performed prior to the stent deployment. Otherwise, the stent will be deployed over a guidewire, under fluoroscopy.
  After, the gastroscopy will go through the esophagus to check for the stent deployment, or any complications.
  An injection of contrast agent will be done to be sure of the correct positioning and that no complications was happened.
  The patient will be kept overnight, with liquid food for 3 days and under PPI until one month after the stent placement.
Device: Stent removal — Six months after implantation, the removal of the stent will be performed. Patient will undergo a first endoscopy under general anesthesia for the placement of a FCSEMS. Then, depending on the importance of the hyperplasia, removal of both stents, under general anesthesia, will be done after 7 to 10 days.

SUMMARY:
A novel stent, called Universal Partially Covered Removable Self-expanding Stent and Anchoring System for the Treatment of Refractory Benign Esophageal Strictures (UAS-RBS) was designed to improve the treatment of benign esophageal refractory strictures with a novel stent. This study aims at evaluating the safety of this new device.

DETAILED DESCRIPTION:
Refractory strictures are defined as benign esophageal strictures who do not achieve acceptable symptom relief despite an intensive dilation schedule. Considering the failure of balloon or mechanical dilation other techniques such as intralesional injection of corticosteroids or stents placement were developed.

Self-expandable metal stents, plastic stents and biodegradable stents are also used in that indication. In a meta-analysis of 18 studies with 444 patients, clinical success was achieved in 41 percent of patients. Stent migration occurred in 29 percent of patients, and adverse events occurred in 21 percent.

A self-expending nitinol stent has been design to reduce the migration risk. The stent is partially covered on both extremities, allowing the formation of small hyperplasia in the middle part of the stent. This design with the inner sheet (usually, when using fully covered stents, the sheet is outside) allows formation of hyperplasia (therefore reducing the risk of migration) but partly controlled by the inner sheet to reduce the risk of lumen occlusion. By this design, the balance between hyperplasia formation to avoid the risk of migration and reducing the risk of lumen occlusion could be entailed stable esophageal calibration.

The UAS-RBS system is a reversible procedure to treat Refractory Benign Esophageal Strictures through stent implantation. Above standard of care monitoring, safety assessment of the procedure and device performance decreases the risk and unforeseen events.

ELIGIBILITY:
Inclusion Criteria:

* Benign Esophageal Refractory Stricture no more than 40 mm in length.
* More than two dilations to at least 16 mm in diameter with symptoms relapse within 6 months.
* Last dilation to 16 mm no more than 6 months before study procedure.
* Dysphagia score of 2 (ability to swallow semi-solid foods), 3 (ability to swallow liquids only) or 4 (unable to swallow liquids) at the time of measurement.
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Stricture within 2 cm of the upper esophageal sphincter.
* Dysphagia related to motility disorder.
* Planned adjuvant radiation therapy post esophagectomy.
* Esophageal stent in place.
* Active erosive esophagitis.
* Sensitivity to any components of the stent or delivery system.
* Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety.
* Currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of all Adverse Device Effects | 6 months
  Serious adverse event (SAE) during the period of stent implantation
Technical stent placement success | Day 0
  Ability to deploy the UAS-RBS in satisfactory position across the stricture
Full deployment of stent | Day 0
  Endoscopic visualization
Technical stent removal success | up to 6 months
  Ability to remove the stent without complications

SECONDARY OUTCOMES:
SAE during the period after stent removal | 6 months post retrieval
Number of re-interventions | within 12 months following stent placement
Change of dysphagia score (Dakkak and Bennett score of Dysphagia) | Baseline and at week 1, month 1, 2, 3, 6, 9, 12 after implantation
Patient's satisfaction with the therapy | week 1, month 1, 2, 3, 6, 9, 12 after implantation
  scored by a visual analog scale (0 worse - 10 best)
Patient's report of pain | before treatment, and at week 1, month 1, 2, 3, 6, 9, 12 after implantation
  scored by a visual analog scale (0 worse - 10 best)
Quality Of Life SF36 questionnaire | before treatment, and at week 1, month 1, 2, 3, 6, 9, 12 after implantation
  SF36

CONTACTS AND LOCATIONS:
Locations (1):
- CUB Hopital erasme, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No